CLINICAL TRIAL: NCT04686279
Title: Safety, PK/PD, Acceptability, and Desirability of a Novel HIV Prevention Douche Among Adolescent Men (DREAM)
Brief Title: Tenofovir Rectal Douche to Prevent HIV Transmission Among Adolescents (ATN DREAM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Emory University (Other); Johns Hopkins University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATN 163
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS; HIV Prevention
Keywords: Tenofovir; Tenofovir Douche
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TFV Medicated Douche (Experimental): Once enrolled, participants will complete a baseline sampling session and then a single dose of study product administration. Post-dose observations and data collection will follow at 1, 6, 24, and 72 hours, using a sparse PK sampling design in which plasma and peripheral blood mononuclear cells (PBMC) are collected at each designated time. Between sampling windows, YMSM will complete a web-survey examining their perceived reactions and comfort using the study douche, factors influencing product use in the future, and comfort with the trial procedures. The survey will be administered after dosing but scheduled not to interfere with other study assessments. Sampling for safety, PK, PD, and acceptability assessments will be collected according to the schedule of events. Phase I Trial participants will complete an in-depth interview as part of their Termination visit.
  Interventions: Drug: Tenofovir Douche

INTERVENTIONS:
Drug: Tenofovir Douche — 660 mg TFV in 125 mL hypo-osmolar solution

SUMMARY:
ATN DREAM is an early phase-1, open label study to examine the safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of a one-dose tenofovir (TFV) medicated douche. The overall goal is to inform the design of an extended safety study of an on-demand and behaviorally congruent TFV douche to confer protection from HIV acquisition in an outpatient pre-RAI context

DETAILED DESCRIPTION:
On demand and behaviorally-congruent forms of HIV pre-exposure prophylaxis (PrEP) have long been demanded by communities at great risk of HIV, especially men who have sex with men (MSM). The DREAM Program is developing a tenofovir (TFV) douche for on demand PrEP use prior to receptive anal intercourse (RAI), given that the vast majority of MSM very commonly douche prior to RAI (behaviorally-congruent). This ATN protocol seeks to ensure the inclusion of adolescent and young adults' (age 15-24 years) perspectives as next generation biomedical prevention, specifically a rectal douche, is being developed for efficacy.

ATN DREAM is an early phase 1, open label study to compare the safety, PK, PD, and acceptability of a TFV-medicated douche. Each participant will undergo a Screening Visit to evaluate eligibility. Baseline Visit will assess pre-dose safety, PK, PD, and behavioral points of reference. Safety, PK, PD, and behavioral readouts are assessed at specified times after the single dose. The TFV douche to be used consists of TFV 660 mg in 125 mL half-normal saline (TFV 5.28 mg/mL). Study objectives including safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of a single TFV douche, are essential to inform the design of an extended safety study of a TFV douche in outpatient pre-RAI contexts. The necessity of extending the testing of new HIV prevention modalities to this proposed adolescent population is motivated by anticipated behavioral differences, not biological ones.

Participant accrual will take approximately 9 months and each participant will be on study for approximately 3 months. Total study duration is about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-24 at Screening
* Cisgender male who has sex with other men
* Willing and able to communicate in English
* Willing and able to provide informed consent to take part in the study
* Participant demonstrates capacity to comprehend, evaluate, reason, and express a choice about their participation in study
* For youth ages 15-17, have parent or caregiver consent to take part in the study
* Willing and able to provide adequate locator information
* Express initial interest in participating in a douching study
* Understand and agree to local HIV/STI reporting requirements
* HIV-1 uninfected at screening as documented by Combo Ag/Ab HIV- 1/HIV-2 immunoassay
* Willingness and availability to attend all study visits, barring unforeseen circumstances
* Per participant report at screening, consensual RAI in prior 6 months
* Live in or around the Baltimore area.
* Willing to abstain from insertion of anything (drug/medication, digits, penis, object, sex toy, or douche) into the anorectum for 72 hours before and after each study visit and 7 days after the biopsy collection.
* Willing to refrain from aspirin, vitamins and herbal supplements, and NSAID use for one week before and after each study biopsy visit
* Agrees not to participate in other research studies involving drugs and/ or medical devices for the study's duration

Exclusion Criteria:

* Participation in research studies involving drugs, medical devices, genital products, or vaccines within 30 days of the Enrollment Visit.
* History of Hepatitis B infection, as documented by positive HBsAg at screening
* ≥ Grade 2 laboratory abnormality at baseline as defined by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 - July 2017, and Addendum 3 (Rectal Grading Tables for Use in Microbicide Studies)
* Self-report as having used TDF 300 mg/FTC 200 mg (Truvada®) or TAF 25 mg/FTC 200 mg (Descovy®) as HIV PrEP or Truvada as PEP within three weeks of dosing visit.
* Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
* At screening or within the past 2 months: participant- reported symptoms and/or clinical or laboratory diagnosis of active rectal infection requiring treatment per current CDC guidelines. Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion. (Note: if an STI apart from HIV is detected, the participant will be referred for treatment and can be retested in 30 days and rescreened once).
* History of an underlying clinically significant cardiac arrhythmia or renal disease (including creatinine clearance <60 mL/min using Cockcroft-Gault equation)
* Serum phosphate < 2.3 mg/dL
* History of significant gastrointestinal bleeding
* Current use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], NSAIDs, or Pradaxa®)
* Use of systemic or anorectal immunomodulatory medications within 4 weeks of enrollment or planned use at any time during study participation
* Per participant report, use of any rectally administered products containing N-9 (including condoms) or investigational products within 4 weeks of enrollment, or planned use of either at any time during study participation
* Known allergic reaction to TFV or other components of the test articles
* Current known HIV-positive partner(s)
* History of recurrent urticaria
* Symptoms suggestive of acute HIV seroconversion at screening and enrollment
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements.
* Presence of substance use (e.g., Cocaine, Marijuana, Opiates, Amphetamines, Methamphetamine, Phencyclidine, Benzodiazepine, Methadone, Barbiturate, Tricyclic Antidepressants, Oxycodone, and Propoxyphene) in one-step urine drug test.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig W Hendrix, MD, Principal Investigator — Johns Hopkins University; Renata Arrington-Sanders, MD, Study Director — Johns Hopkins University; Allison L Agwu, MD, Study Director — Johns Hopkins University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauermeister JA, Arrington-Sanders R, Coleman-Lewis J, Bertagnolli LN, Massih S, Marzinke MA, Fuchs EJ, Zheng R, Anderson T, Addison B, Yang YH, Breakey J, Hoffman J, Bakshi RP, Zak AM, Beselman S, Lin W, Agwu AL, Hightow-Weidman L, Hendrix CW. Safety, Pharmacokinetics, and Acceptability of a Tenofovir Rectal Microbicide Douche Among Young Men Who Have Sex With Men: The DREAM ATN Study (ATN 163). J Infect Dis. 2025 Oct 15;232(4):826-834. doi: 10.1093/infdis/jiaf349. PMID 40578814
- [Derived] Bauermeister JA, Lin W, Webster J, Listerud LL, Burgese T, Agwu A, Lewis JC, Anderson T, Hightow-Weidman L, Hendrix C, Arrington-Sanders R. Assessing the Acceptability of a Tenofovir-Based Rectal Microbicide Douche among Young Men who Have Sex with Men: Results from ATN-DREAM (ATN 163). AIDS Behav. 2025 Oct;29(10):3114-3124. doi: 10.1007/s10461-025-04763-2. Epub 2025 May 29. PMID 40439767

RESULTS

PARTICIPANT FLOW:
Groups:
- TFV Medicated Douche: Once enrolled, participants will complete a baseline sampling session and then a single dose of study product administration. Post-dose observations and data collection will follow at 1, 24, or 72 hours, using a sparse PK sampling design in which plasma and peripheral blood mononuclear cells (PBMC) are collected at each designated time. Between sampling windows, YMSM will complete a web-survey examining their perceived reactions and comfort using the study douche, factors influencing product use in the future, and comfort with the trial procedures. The survey will be administered after dosing but scheduled not to interfere with other study assessments. Sampling for safety, PK, PD, and acceptability assessments will be collected according to the schedule of events. Phase I Trial participants will complete an in-depth interview as part of their Termination visit.
  Tenofovir Douche: 660 mg TFV in 125 mL hypo-osmolar solution
Period: Overall Study
Arm/Group | TFV Medicated Douche
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TFV Medicated Douche
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: Years] | 21 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Body Mass Index [Median (Full Range); unit: kg/m^2] | 27.0 [22.7 to 36.2]

OUTCOME MEASURES:

1. Primary Outcome: Tenofovir Diphosphate (TFV-DP) Concentration
Description: Colonic tissue cell TFV-DP concentrations (femtomoles/million cells) will be measured the study douche administration, based on the individual participant's sampling schedule, on Day 1 (at 1 hour post dose), Day 2 (24 hours post dose), or Day 4 (72 hours post dose).
Time Frame: At 1 hour, 24 hours, or 72 hours after the TFV douche administration
Population: Participants assigned to each sampling schedule (1 hr, 24hr, 72 hr) are included below.
Measure: Median (Full Range); unit: femtomole/million cells
Groups:
- TFV Medicated Douche: Once enrolled, participants will complete a baseline sampling session and then a single dose of study product administration. Post-dose observations and data collection will follow at 1, 24, and 72 hours, using a sparse PK sampling design in which plasma and peripheral blood mononuclear cells (PBMC) are collected at each designated time. Between sampling windows, YMSM will complete a web-survey examining their perceived reactions and comfort using the study douche, factors influencing product use in the future, and comfort with the trial procedures. The survey will be administered after dosing but scheduled not to interfere with other study assessments. Sampling for safety, PK, PD, and acceptability assessments will be collected according to the schedule of events. Phase I Trial participants will complete an in-depth interview as part of their Termination visit.
  Tenofovir Douche: 660 mg TFV in 125 mL hypo-osmolar solution
Arm/Group | TFV Medicated Douche
Number analyzed (Participants) | 8
femtomole/million cells
  1 hour post-dose: number analyzed (Participants) | 4
  1 hour post-dose | 2441 [1033 to 5108]
  24 hours post-dose: number analyzed (Participants) | 3
  24 hours post-dose | 3472 [772 to 9460]
  72 Hours post-dose: number analyzed (Participants) | 1
  72 Hours post-dose | 406 [406 to 406]

2. Primary Outcome: Acceptability of TFV Douche as Assessed by Product Acceptability Questionnaire
Description: Using a 4-point scale (1=Completely Unacceptable; 2=Somewhat Unacceptable; 3=Somewhat Acceptable; 4=Highly Acceptable), participants were asked to answer the following question about their experience with the product: "If a rectal douche like the one you were administered today at the clinic could protect you against HIV, would you consider using this douche?". The endpoint was operationalized as binary, with scores 1 to 2 grouped as "low acceptability" and scores 3 to 4 as "high acceptability".
Time Frame: Following administration of study product, up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | TFV Medicated Douche
Number analyzed (Participants) | 8
Participants
  Low Acceptability | 0
  High Acceptability | 8

3. Primary Outcome: Safety of TFV Douche as Assessed by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events
Description: The safety of a single dose of a TFV douche when applied rectally is measured by the number of ≥Grade 2 adverse events (AEs) as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, and whether AEs are attributed to the study product.
Time Frame: Following administration of study product, up to 7 days
Measure: Number; unit: events
Arm/Group | TFV Medicated Douche
Number analyzed (Participants) | 8
events
  Number of Grade 2 Adverse Events | 3
  Number of Grade 2 AEs attributed to study product | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial (3 months)
Arm/Group | TFV Medicated Douche
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TFV Medicated Douche (N=8)
Nausea (Gastrointestinal disorders) | 1 (1)
Type I Diabetes (Metabolism and nutrition disorders) | 2 (3) — Grade 2 Fasting Glucose. Not related to study given participant underlying condition (Type 1 Diabetes)
Polyp (Gastrointestinal disorders) | 1 (1) — Detection of sessile polyps detected during a flexible sigmoidoscopy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT04686279/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04686279/ICF_001.pdf